CLINICAL TRIAL: NCT04394351
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of Dupilumab in Pediatric Patients With Active Eosinophilic Esophagitis
Brief Title: Study to Investigate the Efficacy and Safety of Dupilumab in Pediatric Patients With Active Eosinophilic Esophagitis (EoE)
Acronym: EoE KIDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R668-EE-1877; 2019-003078-24 (EudraCT Number)
Record Dates: First submitted 2020-05-07; First posted 2020-05-19 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Eosinophilic Esophagitis (EoE)
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A - High Dose (Experimental): Part A consists of a 16-week double-blind treatment period. Patients will be randomized to receive dupilumab or placebo subcutaneous (SC) administration at tiered dosing regimens based on body weight
  Interventions: Drug: Dupilumab; Drug: Matching Placebo
- Part A - Low Dose (Experimental): Part A consists of a 16-week double-blind treatment period. Patients will be randomized to receive dupilumab or placebo subcutaneous (SC) administration at tiered dosing regimens based on body weight
  Interventions: Drug: Dupilumab; Drug: Matching Placebo
- Part B - High Dose (Experimental): Part B consists of a 36-week extended active treatment period. All patients to receive subcutaneous (SC) administration at tiered dosing regimens based on body weight
  Interventions: Drug: Dupilumab; Drug: Matching Placebo
- Part B - Low Dose (Experimental): Part B consists of a 36-week extended active treatment period. All patients to receive subcutaneous (SC) administration at tiered dosing regimens based on body weight
  Interventions: Drug: Dupilumab; Drug: Matching Placebo
- Part C - High Dose (Experimental): Part C consists of up to 108-week open-label extension period. All patients will receive higher exposure dupilumab subcutaneous (SC) administration at tiered dosing regimens based on body weight. No matching placebo administered in Part C.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Single-use, prefilled syringe
  Other Names: •DUPIXENT; •REGN668; •SAR231893
Drug: Matching Placebo — Matching formulation and regimen (depending on the weight tier) as dupilumab without the active substance
  Arms: Part A - High Dose; Part A - Low Dose; Part B - High Dose; Part B - Low Dose

SUMMARY:
The Primary objective is to demonstrate the efficacy of dupilumab treatment compared with placebo in pediatric patients with active eosinophilic esophagitis (EoE) based on histologic improvement meeting validated histologic criteria.

The Secondary objectives are:

* To demonstrate the efficacy of dupilumab compared to placebo in pediatric patients with active EoE after 16 weeks of treatment as assessed by endoscopic visual measurements of disease activity using the Eosinophilic Esophagitis-Endoscopic Reference Score (EoE-EREFS) and histologic abnormalities as measured by the EoE Histology Scoring System (EoE-HSS)
* To evaluate the safety, tolerability, and immunogenicity of dupilumab treatment for up to 16 weeks in pediatric patients with active EoE
* To evaluate the effects of dupilumab on transcriptomic signatures associated with EoE and type 2 inflammation
* To study the effects of dupilumab on the type 2 inflammation gene expression signature
* To evaluate the concentration-time profile of functional dupilumab in serum in this population
* To assess efficacy of long-term (up to 160 weeks) dupilumab treatment
* To assess the impact of dupilumab treatment on changes in weight and growth during the extended active period and open-label extension period of the study
* To assess safety, tolerability, and immunogenicity of long-term (up to 160 weeks) dupilumab treatment
* To evaluate the impact of dupilumab treatment on EoE signs and symptoms

DETAILED DESCRIPTION:
This is a 3-part study:

* Part A: Double-blind 16-week treatment period
* Part B: 36-week extended active treatment period
* Part C: Up to108 weeks open-label extension period

ELIGIBILITY:
Key Inclusion Criteria:

1. A documented diagnosis of eosinophilic esophagitis (EoE)
2. Baseline endoscopic biopsies with a demonstration on central reading of intraepithelial eosinophilic infiltration

Key Exclusion Criteria:

1. Body weight <5 kg or ≥60 kg at screening
2. Other causes of esophageal eosinophilia
3. Active Helicobacter pylori
4. History of Crohn's disease, ulcerative colitis, celiac disease, or prior esophageal surgery
5. Any esophageal stricture unable to be passed with a standard, diagnostic, upper endoscope or any critical esophageal stricture that requires dilation at screening
6. Treatment with swallowed topical corticosteroids within 8 weeks prior to baseline standard of care endoscopy
7. History of bleeding disorders or esophageal varices that, in the opinion of the investigator, would put the patient at undue risk for significant complications from an endoscopy procedure
8. Active parasitic infection or suspected parasitic infection
9. Known or suspected immunodeficiency disorder

Key Exclusion for Patients Re-Entering the Study (for Entry into Part C, as defined in protocol):

1. Patients who are ≥12 years old, weigh ≥40 kg (or minimum weight for which dupilumab is approved for EoE), and dupilumab is commercially available for the treatment of EoE in their country
2. Patients who, during their previous participation in this clinical trial, developed an SAE and/or AE deemed related to dupilumab, which in the opinion of the investigator or of the medical monitor could indicate that continued treatment with dupilumab may present an unreasonable risk for the patient
3. Patients who did not undergo endoscopy with biopsies at week 16 and/or week 52 or prior to receiving rescue treatment Note: If the endoscopy with biopsies could not occur due to COVID-19 restrictions and rescue treatment was needed to be initiated without delay, these patients will be eligible to participate in Part C
4. Patients who became pregnant during their previous participation in this dupilumab clinical trial
5. Patients who, during their previous participation in this trial, were prematurely withdrawn because of a protocol violation, poor compliance, or inability to complete required study assessments

NOTE: Other protocol defined inclusion/exclusion criteria apply

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2024-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (22):
- United States (21):
  - Regeneron Study Site, Phoenix, Arizona
  - Regeneron Study Site, Little Rock, Arkansas
  - Regeneron Study Site, Los Angeles, California
  - Regeneron Study Site, San Francisco, California
  - Regeneron Study Site, Aurora, Colorado
  - Regeneron Study Site, St. Petersburg, Florida
  - Regeneron Study Site, Atlanta, Georgia
  - Regeneron Study Site, Chicago, Illinois
  - Regeneron Study Site, Indianapolis, Indiana
  - Regeneron Study Site, Iowa City, Iowa
  - Regeneron Study Site, Boston, Massachusetts
  - Regeneron Study Site, Lincoln, Nebraska
  - Regeneron Study Site, New York, New York
  - Regeneron Study Site, Chapel Hill, North Carolina
  - Regeneron Study Site, Cincinnati, Ohio
  - Regeneron Study Site, Cleveland, Ohio
  - Regeneron Study Site, Philadelphia, Pennsylvania
  - Regeneron Study Site, Dallas, Texas
  - Regeneron Study Site, Fort Worth, Texas
  - Regeneron Study Site, Houston, Texas
  - Regeneron Study Site, Milwaukee, Wisconsin
- Regeneron Study Site, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

REFERENCES:
- [Derived] Chehade M, Dellon ES, Spergel JM, Collins MH, Rothenberg ME, Pesek RD, Hirano I, Liu R, Laws E, Mortensen E, Martincova R, Shabbir A, McCann E, Kamal MA, Kosloski MP, Hamilton JD, Samuely C, Lim WK, Wipperman MF, Farrell A, Patel N, Yancopoulos GD, Glotfelty L, Maloney J. Dupilumab for Eosinophilic Esophagitis in Patients 1 to 11 Years of Age. N Engl J Med. 2024 Jun 27;390(24):2239-2251. doi: 10.1056/NEJMoa2312282. PMID 38924731

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of 3 parts: Part A (double-blind 16-week treatment period), Part B (36-week extended active treatment period) and Part C (open-label extension period of up to 108 weeks).
Groups:
- Part A: Pooled Placebo (Placebo): Participants who received subcutaneous (SC) injection of placebo matched to higher exposure dupilumab or lower exposure dupilumab in Part A. Lower exposure dupilumab regimen were exposures approximating those in adolescents and adults receiving 300 mg dupilumab Q2W). Higher exposure dupilumab regimen were exposures approximating those in adolescents and adults receiving 300 mg dupilumab QW.
- Part A: Dupilumab Low Dose: Participants received subcutaneous (SC) injection of lower exposure dupilumab in Part A. Lower exposure dupilumab regimen were exposures approximating those in adolescents and adults receiving 300 mg dupilumab Q2W
- Part A: Dupilumab High Dose: Participants received subcutaneous (SC) injection of higher exposure dupilumab in Part A. Higher exposure dupilumab regimen were exposures approximating those in adolescents and adults receiving 300 mg dupilumab QW
- Part B: Placebo to Dupilumab Low Dose: Participants who received subcutaneous (SC) injection of placebo in Part A and received lower exposure dupilumab in Part B. Lower exposure dupilumab regimen were exposures approximating those in adolescents and adults receiving 300 mg dupilumab Q2W
- Part B: Placebo to Dupilumab High Dose: Participants who received subcutaneous (SC) injection of placebo in Part A and received higher exposure dupilumab in Part B. Higher exposure dupilumab regimen were exposures approximating those in adolescents and adults receiving 300 mg dupilumab QW
- Part B: Dupilumab Low Dose to Dupilumab Low Dose: Participants received subcutaneous (SC) injection of lower exposure dupilumab in Parts A and B. Lower exposure dupilumab regimen were exposures approximating those in adolescents and adults receiving 300 mg dupilumab Q2W)
- Part B: Dupilumab High Dose to Dupilumab High Dose: Participants received subcutaneous (SC) injection of higher exposure dupilumab in Parts A and B. Higher exposure dupilumab regimen were exposures approximating those in adolescents and adults receiving 300 mg dupilumab QW.
- Part C: Dupilumab: Participants who completed Part A and B were eligible to enroll in Part C and receive Dupilumab extended active treatment
Period: Part A (16 Weeks)
Arm/Group | Part A: Pooled Placebo (Placebo) | Part A: Dupilumab Low Dose | Part A: Dupilumab High Dose | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose | Part C: Dupilumab
Started | 34 | 31 | 37 | 0 | 0 | 0 | 0 | 0
Completed | 33 | 29 | 37 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (36 Weeks)
Arm/Group | Part A: Pooled Placebo (Placebo) | Part A: Dupilumab Low Dose | Part A: Dupilumab High Dose | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose | Part C: Dupilumab
Started | 0 | 0 | 0 | 14 | 18 | 29 | 37 | 0
Completed | 0 | 0 | 0 | 14 | 18 | 29 | 36 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Part C: (Up to Wk108+12Wk Follow-up)
Arm/Group | Part A: Pooled Placebo (Placebo) | Part A: Dupilumab Low Dose | Part A: Dupilumab High Dose | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose | Part C: Dupilumab
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 61
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 53
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 32

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Part A full analysis set (FAS) which included all randomized participants in Part A.
Groups:
- Part A: Pooled Placebo: Participants who received subcutaneous (SC) injection of placebo matched to higher exposure dupilumab or lower exposure dupilumab in Part A. Lower exposure dupilumab regimen were exposures approximating those in adolescents and adults receiving 300 mg dupilumab Q2W). Higher exposure dupilumab regimen were exposures approximating those in adolescents and adults receiving 300 mg dupilumab QW.
- Total: Total of all reporting groups
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab Low Dose | Part A: Dupilumab High Dose | Total
Number analyzed (Participants) | 34 | 31 | 37 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.2 (3.03) | 7.2 (3.07) | 6.8 (3.11) | 7.1 (3.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 9 | 24
  Male | 25 | 25 | 28 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 7
  Not Hispanic or Latino | 30 | 29 | 33 | 92
  Unknown or Not Reported | 1 | 0 | 2 | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 30 | 22 | 32 | 84
  Black or African American | 3 | 4 | 4 | 11
  Asian | 0 | 1 | 1 | 2
  Other | 1 | 4 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Part A: Percentage of Participants Achieving Peak Esophageal Intraepithelial Eosinophil Count of Less Than or Equal to (≤) 6 Eosinophils/High Power Field (Eos/Hpf) at Week 16
Description: Peak esophageal intraepithelial eosinophil count was measured from esophageal biopsies. A total of at least 9 mucosal pinch biopsies were collected from 3 esophageal regions: 3 proximal, 3 mid, and 3 distal. The peak esophageal intraepithelial eosinophil count at each visit was the maximum of the quantities of eosinophils in the most inflamed hpfs across the 3 regions. If the quantity of eosinophils was missing for 1 or 2 esophageal regions, the peak eosinophil count was the maximum of the quantities of eosinophils from the region(s) where eosinophil quantities were available.
Time Frame: At Week 16
Population: Analysis was performed on Part A FAS which included all randomized participants in Part A.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part A: Dupilumab Low Dose: Participants received subcutaneous (SC) injection of lower exposure dupilumab in Part A. Lower exposure dupilumab regimen were exposures approximating those in adolescents and adults receiving 300 mg dupilumab Q2W)
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 34 | 37 | 31
percentage of participants | 2.9 [0.07 to 15.33] | 67.6 [50.21 to 81.99] | 58.1 [39.08 to 75.45]
Statistical Analysis 1: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab High Dose; Part A: Dupilumab High Dose versus Part A: Pooled Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; p-value was derived by Cochran-Mantel-Haenszel (CMH) test stratified by baseline weight group; Odds Ratio (OR) = 53.8, 95% CI 2-sided [7.37 to 392.82] — Odds ratio and corresponding Confidence Interval (CI) are based on CMH test stratified by baseline weight group
Statistical Analysis 2: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab Low Dose; Part A: Dupilumab Low Dose versus Part A: Pooled Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; p-value was derived by CMH test stratified by baseline weight group; Odds Ratio (OR) = 46.7, 95% CI 2-sided [5.47 to 399.54] — Odds ratio and corresponding CI are based on CMH test stratified by baseline weight group

2. Secondary Outcome: Part A: Percentage of Participants Achieving Peak Esophageal Intraepithelial Eosinophil Count of <15 Eosinophils/High Power Field at Week 16
Description: as for outcome 1
Time Frame: At Week 16
Population: Analysis was performed on Part A FAS which included all randomized participants in Part A.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 34 | 37 | 31
percentage of participants | 2.9 [0.07 to 15.33] | 83.8 [67.99 to 93.81] | 67.7 [48.63 to 83.32]
Statistical Analysis 1: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab High Dose; Part A: Dupilumab High Dose versus Part A: Pooled Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; p-value was derived by CMH test stratified by baseline weight group; Odds Ratio (OR) = 178.0, 95% CI 2-sided [18.84 to 1682.4] — Odds ratio and corresponding CI are based on CMH test stratified by baseline weight group
Statistical Analysis 2: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab Low Dose; Part A: Dupilumab Low Dose versus Part A: Pooled Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value is not adjusted for multiple comparisons; p-value was derived by CMH test stratified by baseline weight group; Odds Ratio (OR) = 55.3, 95% CI 2-sided [7.45 to 410.23] — Odds ratio and corresponding CI are based on CMH test stratified by baseline weight group

3. Secondary Outcome: Part A: Percent Change From Baseline in Peak Esophageal Intraepithelial Eosinophil Count at Week 16
Description: Peak esophageal intraepithelial eosinophil count was measured from esophageal biopsies. A total of at least 9 mucosal pinch biopsies were collected from 3 esophageal regions: 3 proximal, 3 mid, and 3 distal. The peak esophageal intraepithelial eosinophil count at each visit was the maximum of the quantities of eosinophils in the most inflamed hpfs across the 3 regions. If the quantity of eosinophils was missing for 1 or 2 esophageal regions, the peak eosinophil count was the maximum of the quantities of eosinophils from the region(s) where eosinophil quantities were available. Least squared (LS) mean and standard error (SE) from analysis of covariance (ANCOVA) model with Baseline measurement as covariate and the treatment, baseline weight group strata as fixed factors.
Time Frame: Baseline, Week 16
Population: Analysis was performed on Part A FAS which included all randomized participants in Part A.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 34 | 37 | 31
percent change | 20.98 (12.23) | -86.09 (11.84) | -77.93 (12.89)
Statistical Analysis 1: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab High Dose; Part A: Dupilumab High Dose versus Part A: Pooled Placebo; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = -107.07, 95% CI 2-sided [-139.249 to -74.900] — CI was based on treatment difference (Dupilumab group vs. placebo) of the LS mean change using ANCOVA model with baseline measurement as covariate and the treatment, baseline weight group strata as fixed factors
Statistical Analysis 2: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab Low Dose; Part A: Dupilumab Low Dose versus Part A: Pooled Placebo; Test type: Superiority; p < 0.0001, ANCOVA — P-value is not adjusted for multiple comparisons; LS mean difference = -98.92, 95% CI 2-sided [-132.463 to -65.370] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Part A: Change From Baseline in Mean Eosinophilic Esophagitis Histology Scoring System (EoE-HSS) Grade Score at Week 16
Description: EoE-HSS is a validated histologic scoring system that measures other histological abnormalities in addition to density of eosinophilic infiltration. Severity (grade) and extent (stage) of abnormalities will be scored using a 4-point scale (0 normal; 3 maximum change). Higher total score indicated greater severity & extent of histological abnormalities. For each of 3 esophageal regions (proximal, mid, and distal), the ratio of the sum of assigned score for each evaluated feature divided by maximum possible score (maximum value is 24) was calculated. The mean grade scores summed over the 3 regions was the final score used in primary analysis, the mean grade score ranged from 0 to 3, with higher score indicating more severe.
Time Frame: Baseline, Week 16
Population: Analysis was performed on Part A FAS which included all randomized participants in Part A.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 34 | 37 | 31
Score on a scale | 0.023 (0.0498) | -0.879 (0.0481) | -0.757 (0.0524)
Statistical Analysis 1: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab High Dose; Part A: Dupilumab High Dose versus Part A: Pooled Placebo; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = -0.902, 95% CI 2-sided [-1.0325 to -0.7714] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab Low Dose; Part A: Dupilumab Low Dose versus Part A: Pooled Placebo; Test type: Superiority; p < 0.0001, ANCOVA — P-value is not adjusted for multiple comparisons; LS mean difference = -0.780, 95% CI 2-sided [-0.9170 to -0.6440] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Part A: Change From Baseline in Mean Eosinophilic Esophagitis Histology Scoring System (EoE-HSS) Stage Score at Week 16
Description: EoE-HSS is a validated histologic scoring system that measures other histological abnormalities in addition to density of eosinophilic infiltration. Severity (grade) and extent (stage) of abnormalities will be scored using a 4-point scale (0 normal; 3 maximum change). Higher total score indicated greater severity & extent of histological abnormalities. For each of 3 esophageal regions (proximal, mid, and distal), the ratio of the sum of assigned score for each evaluated feature divided by maximum possible score (maximum value is 24) was calculated. The mean stage scores summed over the 3 regions was the final score used in primary analysis, the mean stage score ranged from 0 to 3, with higher score indicating more severe.
Time Frame: Baseline, Week 16
Population: Analysis was performed on Part A FAS which included all randomized participants in Part A.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 34 | 37 | 31
Score on a scale | 0.048 (0.0482) | -0.835 (0.0466) | -0.721 (0.0507)
Statistical Analysis 1: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab High Dose; Part A: Dupilumab High Dose versus Part A: Pooled Placebo; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = -0.883, 95% CI 2-sided [-1.0095 to -0.7568] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab Low Dose; Part A: Dupilumab Low Dose versus Part A: Pooled Placebo; Test type: Superiority; p < 0.0001, ANCOVA — P-value is not adjusted for multiple comparisons; LS mean difference = -0.769, 95% CI 2-sided [-0.9013 to -0.6362] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Part A: Normalized Enrichment Score (NES) for the Relative Change From Baseline in the Type 2 Inflammation Signature (T2INF) at Week 16
Description: A Normalized Enrichment Score (NES) is a way to generate a single numerical value to represent a complex gene expression signature. Changes in NES score represented the overall changes in the expression of that molecular phenotype. The NESs calculated for T2INF reflect the expression at Week 16 relative to Baseline of the pre-specified gene set as a way to evaluate normalization of type 2 inflammation with treatment. For each subject, an NES of 0 indicates no change from baseline, a negative score shows a reduction in disease score (more like normal) and positive score shows worsening (more active disease). NES does not have a minimum/maximum score.
Time Frame: Baseline, Week 16
Population: Analysis was performed on Part A FAS which included all randomized participants in Part A. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 21 | 24 | 15
Score on a scale | 0.34 [-1.84 to 1.65] | -1.895 [-2.03 to -1.61] | -1.930 [-2.00 to -1.39]
Statistical Analysis 1: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab High Dose; Part A: Dupilumab High Dose versus Part A: Pooled Placebo; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test; Hodges-Lehmann estimator = -2.220, 95% CI 2-sided [-2.4400 to -1.9500] — Median Difference is Dupilumab minus Placebo
Statistical Analysis 2: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab Low Dose; Part A: Dupilumab Low Dose versus Part A: Pooled Placebo; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test — P-value is not adjusted for multiple comparisons; Hodges-Lehmann estimator = -2.190, 95% CI 2-sided [-2.4500 to -1.8200] — Median Difference is Dupilumab minus Placebo

7. Secondary Outcome: Part A: Normalized Enrichment Score (NES) for the Relative Change From Baseline in the Eosinophilic Esophagitis (EoE) Diagnostic Panel (EDP) at Week 16
Description: A Normalized Enrichment Score (NES) is a way to generate a single numerical value to represent a complex gene expression signature. Changes in NES score represented the overall changes in the expression of that molecular phenotype. The NESs calculated for the EDP reflect the expression at Week 16 relative to Baseline of a gene set that is differentially expressed between esophageal biopsies from EoE participants compared to healthy controls as a way to evaluate normalization of the molecular pathology. For each subject, an NES of 0 indicates no change from baseline, a negative score shows a reduction in disease score (more like normal) and positive score shows worsening (more active disease). NES does not have minimum/maximum score.
Time Frame: Baseline, Week 16
Population: as for outcome 6
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 21 | 24 | 15
Score on a scale | 0.180 [-2.53 to 2.39] | -2.630 [-2.85 to -2.25] | -2.710 [-2.84 to -0.80]
Statistical Analysis 1: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab High Dose; Part A: Dupilumab High Dose versus Part A: Pooled Placebo; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test; Hodges-Lehmann estimator = -2.840, 95% CI 2-sided [-3.3500 to -1.9600] — Median Difference is Dupilumab minus Placebo
Statistical Analysis 2: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab Low Dose; Part A: Dupilumab Low Dose versus Part A: Pooled Placebo; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test — P-value is not adjusted for multiple comparisons; Hodges-Lehmann estimator = -2.700, 95% CI 2-sided [-3.3100 to -1.6200] — Median Difference is Dupilumab minus Placebo

8. Secondary Outcome: Part A: Absolute Change From Baseline in EoE Endoscopic Reference Total Score (EoE-EREFS) at Week 16
Description: The EoE-EREFS is a validated endoscopic scoring system for inflammatory and remodeling features of EoE including edema, rings, exudates, furrows, and stricture. The score was assessed in the proximal and distal esophageal regions with each region scored from 0 to 9 with total scores ranging from 0 to 18. Higher scores indicate worse endoscopic inflammatory and remodeling findings.
Time Frame: Baseline, Week 16
Population: Analysis was performed on Part A FAS which included all randomized participants in Part A.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 34 | 37 | 31
score on a scale | 0.3 (0.45) | -3.5 (0.42) | -3.0 (0.48)
Statistical Analysis 1: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab High Dose; Part A: Dupilumab High Dose versus Part A: Pooled Placebo; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = -3.8, 95% CI 2-sided [-4.94 to -2.63] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab Low Dose; Part A: Dupilumab Low Dose versus Part A: Pooled Placebo; Test type: Superiority; p < 0.0001, ANCOVA — P-value is not adjusted for multiple comparisons; LS mean difference = -3.3, 95% CI 2-sided [-4.59 to -2.10] — [estimate comment as in outcome 3, analysis 1]

9. Secondary Outcome: Part A: Change From Baseline in the Proportion of Days With 1 or More EoE Signs as Measured by Pediatric EoE Sign/Symptom Questionnaire - Caregiver Version (PESQ-C) at Week 16 (for Participants Aged ≥1 to <12 Years)
Description: PESQ-C is a novel, observer-reported outcome measure intended to be completed independently by caregivers of all pediatric EoE participants in the study. PESQ-C measures the signs of EoE observed by the caregiver, including stomach pain, heartburn, acid reflux, regurgitation, vomiting, food refusal, and trouble swallowing food. Data from a 14-day period preceding the baseline visit and a 14-day period preceding week 16 will be used to calculate the proportion of days with 1 or more EoE symptoms.
Time Frame: Baseline, Week 16
Population: Analysis was performed on Part A FAS which included all randomized participants in Part A.
Measure: Least Squares Mean (Standard Error); unit: proportion of days
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 34 | 37 | 31
proportion of days | -0.17 (0.054) | -0.28 (0.052) | -0.18 (0.060)
Statistical Analysis 1: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab High Dose; Part A: Dupilumab High Dose versus Part A: Pooled Placebo; Test type: Superiority; p = 0.1526, ANCOVA; LS mean difference = -0.10, 95% CI 2-sided [-0.244 to 0.038] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab Low Dose; Part A: Dupilumab Low Dose versus Part A: Pooled Placebo; Test type: Superiority; p = 0.9533, ANCOVA — P-value is not adjusted for multiple comparisons; LS mean difference = -0.00, 95% CI 2-sided [-0.155 to 0.146] — [estimate comment as in outcome 3, analysis 1]

10. Secondary Outcome: Part A: Number of Sign-free Days During the 14-day Period Preceding Week 16 as Measured by the PESQ-C (for Participants Aged ≥1 to <12 Years)
Description: PESQ-C is a novel, observer-reported outcome measure intended to be completed independently by caregivers of all pediatric EoE participants in the study. The PESQ-C measures the signs of EoE observed by the caregiver, including stomach pain, heartburn, acid reflux, regurgitation, vomiting, food refusal, and trouble swallowing food. WOCF approach was used for imputing the missing data due to rescue treatment/AE/lack of efficacy, and the multiple imputations approach was used for the missing data due to other reasons. LS mean SE derived from ANCOVA model.
Time Frame: Week 16
Population: Analysis was performed on Part A FAS which included all randomized participants in Part A.
Measure: Least Squares Mean (Standard Error); unit: sign-free days
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 34 | 37 | 31
sign-free days | 8.93 (0.756) | 10.38 (0.735) | 8.93 (0.840)
Statistical Analysis 1: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab High Dose; Part A: Dupilumab High Dose versus Part A: Pooled Placebo; Test type: Superiority; p = 0.1507, ANCOVA — P-value is not adjusted for multiple comparisons; LS mean difference = 1.45, 95% CI 2-sided [-0.527 to 3.422] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab Low Dose; Part A: Dupilumab Low Dose versus Part A: Pooled Placebo; Test type: Superiority; p = 0.9965, ANCOVA — P-value is not adjusted for multiple comparisons; LS mean difference = 0.00, 95% CI 2-sided [-2.107 to 2.117] — [estimate comment as in outcome 3, analysis 1]

11. Secondary Outcome: Part A: Change From Baseline in the Proportion of Total Segments Within a Day (Night, Morning, Afternoon, Evening) With 1 or More EoE Signs as Measured by the PESQ-C at Week 16
Description: PESQ-C is a novel, observer-reported outcome measure intended to be completed independently by caregivers of all pediatric EoE participants in the study. The PESQ-C measured the occurrence of signs of EoE and was completed once daily via an electronic diary. Data from a 14-day period preceding the baseline visit and a 14-day period preceding week 16 will be used to calculate the total time segments within a day (night, morning, afternoon, evening) with 1 or more EoE symptoms.
Time Frame: Baseline, Week 16
Population: Analysis was performed on Part A FAS which included all randomized participants in Part A.
Measure: Least Squares Mean (Standard Error); unit: proportion of segments
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 34 | 37 | 31
proportion of segments | -0.11 (0.032) | -0.16 (0.031) | -0.09 (0.036)
Statistical Analysis 1: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab High Dose; Part A: Dupilumab High Dose versus Part A: Pooled Placebo; Test type: Superiority; p = 0.2064, ANCOVA — P-value is not adjusted for multiple comparisons; LS mean difference = -0.05, 95% CI 2-sided [-0.139 to 0.030] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab Low Dose; Part A: Dupilumab Low Dose versus Part A: Pooled Placebo; Test type: Superiority; p = 0.6361, ANCOVA — P-value is not adjusted for multiple comparisons; LS mean difference = 0.02, 95% CI 2-sided [-0.069 to 0.112] — [estimate comment as in outcome 3, analysis 1]

12. Secondary Outcome: Part A: Change From Baseline in the Proportion of Days With 1 or More EoE Signs by Pediatric EoE Sign/Symptom Questionnaire - Participant Version (PESQ-P) (for Participants Aged ≥8 to <12 Years) at Week 16
Description: The PESQ-P was a participant-reported outcome measure intended to be completed independently by participants ≥8 to <12 years of age. The PESQ-P measured occurrence of signs of EoE and was completed once daily via an electronic diary. Data from a 14-day period preceding the baseline visit and a 14-day period preceding week 16 will be used to calculate the proportion of days with 1 or more EoE symptoms.
Time Frame: Baseline, Week 16
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: proportion of days
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 17 | 17 | 19
proportion of days | -0.26 (0.068) | -0.13 (0.077) | -0.16 (0.067)
Statistical Analysis 1: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab High Dose; Part A: Dupilumab High Dose versus Part A: Pooled Placebo; Test type: Superiority; p = 0.2086, ANCOVA — P-value is not adjusted for multiple comparisons; LS mean difference = 0.13, 95% CI 2-sided [-0.072 to 0.330] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab Low Dose; Part A: Dupilumab Low Dose versus Part A: Pooled Placebo; Test type: Superiority; p = 0.2975, ANCOVA — P-value is not adjusted for multiple comparisons; LS mean difference = 0.10, 95% CI 2-sided [-0.088 to 0.286] — [estimate comment as in outcome 3, analysis 1]

13. Secondary Outcome: Part A: Number of Symptom-free Days During the 14-day Period Preceding Week 16 as Measured by the PESQ-P (for Participants Aged ≥8 to <12 Years)
Description: The PESQ-P was a participant-reported outcome measure intended to be completed independently by EoE participants ≥8 to <12 years of age. The PESQ-P measures the signs of EoE, including stomach pain, heartburn, acid reflux, regurgitation, vomiting, food refusal, and trouble swallowing food. The PESQ-P score was calculated based on the daily responses over a 14-day period (i.e., the 14 days prior to the baseline visit and the week 16 visit). The score ranges from 0 to 1. WOCF approach was used for imputing the missing data due to rescue treatment/AE/lack of efficacy, and the multiple imputations approach was used for the missing data due to other reasons. LS Mean SE from ANCOVA.
Time Frame: Week 16
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: sign-free days
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 17 | 17 | 19
sign-free days | 10.49 (0.953) | 8.69 (1.081) | 9.13 (0.936)
Statistical Analysis 1: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab High Dose; Part A: Dupilumab High Dose versus Part A: Pooled Placebo; Test type: Superiority; p = 0.2085, ANCOVA — P-value is not adjusted for multiple comparisons; LS mean difference = -1.80, 95% CI 2-sided [-4.615 to 1.007] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab Low Dose; Part A: Dupilumab Low Dose versus Part A: Pooled Placebo; Test type: Superiority; p = 0.3098, ANCOVA — P-value is not adjusted for multiple comparisons; LS mean difference = -1.36, 95% CI 2-sided [-3.972 to 1.260] — [estimate comment as in outcome 3, analysis 1]

14. Secondary Outcome: Part A: Change From Baseline in the Proportion of Total Segments Within a Day (Night, Morning, Afternoon, Evening) With 1 or More EoE Signs as Measured by the PESQ-P (for Participants Aged ≥8 to <12 Years) at Week 16
Description: The PESQ-P was a participant-reported outcome measure intended to be completed independently by EoE participants ≥8 to <12 years of age. The PESQ-P measured the occurrence of signs of EoE and was completed once daily via an electronic diary. Data from a 14-day period preceding the baseline visit and a 14-day period preceding week 16 will be used to calculate the total time segments within a day (night, morning, afternoon, evening) with 1 or more EoE symptoms.
Time Frame: Baseline, Week 16
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: proportion of segments
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 17 | 17 | 19
proportion of segments | -0.15 (0.040) | -0.08 (0.045) | -0.08 (0.039)
Statistical Analysis 1: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab High Dose; Part A: Dupilumab High Dose versus Part A: Pooled Placebo; Test type: Superiority; p = 0.2360, ANCOVA — P-value is not adjusted for multiple comparisons; LS mean difference = 0.07, 95% CI 2-sided [-0.046 to 0.186] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Part A: Pooled Placebo vs Part A: Dupilumab Low Dose; Part A: Dupilumab Low Dose versus Part A: Pooled Placebo; Test type: Superiority; p = 0.1939, ANCOVA — P-value is not adjusted for multiple comparisons; LS mean difference = 0.07, 95% CI 2-sided [-0.037 to 0.181] — [estimate comment as in outcome 3, analysis 1]

15. Secondary Outcome: Part A: Change From Baseline in Total Score as Measured by the Pediatric Eosinophilic Esophagitis Symptom Score (PEESS) Version 2.0 Caregiver Version (PEESSv2.0-C) at Week 16
Description: The PEESSv2.0-C is a caregiver-reported outcome measure that assesses the frequency and severity of EoE symptoms among pediatric participants. The PEESSv2.0-C consists of 20 items and has a one-month recall period. Each item had a 0-4 scale, which was transformed to 0-100 as follows: 0 = 0, 1 = 25, 2 = 50, 3 = 75, 4 = 100. The mean total PEESSv2.0 score was computed as the sum of all the item scores over the number of items answered. The total PEESSv2.0-C score ranges from 0 to 100 where higher scores indicate greater symptom burden among pediatric EoE participants. Values after first rescue treatment use were set to missing (censoring). WOCF approach was used for imputing the missing data due to rescue treatment/AE/lack of efficacy, and the MI approach was used for the missing data due to other reasons. LS mean SE from ANCOVA model.
Time Frame: Baseline, Week 16
Population: Analysis was performed on Part A FAS which included all randomized participants in Part A.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 34 | 37 | 31
score on a scale | -11.83 (2.909) | -19.86 (2.577) | -10.10 (2.785)

16. Secondary Outcome: Part A: Concentration of Functional Dupilumab in Serum at Baseline, Week 4 and 16
Description: Concentration of functional dupilumab in serum at Baseline, Week 4 and 16 was reported in this outcome measure.
Time Frame: Baseline, Week 4 and 16
Population: Analysis was performed on pharmacokinetic analysis set (PKAS) that includes all participants who received any study drug and had at least 1 non-missing result following the first dose of study drug. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 36 | 28
milligrams per liter (mg/L)
  Baseline | 0 (0) | 0 (0)
  Week 4: number analyzed (Participants) | 36 | 26
  Week 4 | 75.7 (25.7) | 40.6 (11.2)
  Week 16: number analyzed (Participants) | 30 | 26
  Week 16 | 163 (60.8) | 86.0 (29.2)

17. Secondary Outcome: Part B: Percentage of Participants Achieving Peak Esophageal Intraepithelial Eosinophil Count of ≤6 Eosinophils/High Power Field at Week 52
Description: as for outcome 1
Time Frame: At Week 52
Population: Analysis was performed on Part B safety analysis set (SAF) which included all participants who received at least 1 dose of Part B study drug. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Groups:
- Part B: Placebo to Dupilumab Low Dose: Participants who received subcutaneous (SC) injection of placebo in Part A and received lower exposure dupilumab in Part B. Lower exposure dupilumab regimen were exposures approximating those in adolescents and adults receiving 300 mg dupilumab Q2W)
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 14 | 17 | 29 | 35
percentage of participants | 92.9 | 52.9 | 65.5 | 62.9

18. Secondary Outcome: Part B: Percentage of Participants Achieving Peak Esophageal Intraepithelial Eosinophil Count of <15 Eosinophils/High Power Field at Week 52
Description: as for outcome 1
Time Frame: At Week 52
Population: Analysis was performed on Part B SAF which included all participants who received at least 1 dose of Part B study drug. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 14 | 17 | 29 | 35
percentage of participants | 92.9 | 64.7 | 69.0 | 85.7

19. Secondary Outcome: Part B: Percent Change From Baseline in Peak Esophageal Intraepithelial Eosinophil Count at Week 52
Description: as for outcome 1
Time Frame: Baseline, Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 14 | 17 | 29 | 35
percent change | -92.72 (19.229) | -76.83 (41.228) | -85.41 (22.851) | -90.97 (14.482)

20. Secondary Outcome: Part B: Change From Baseline in Mean Eosinophilic Esophagitis Histology Scoring System (EoE-HSS) Grade Score at Week 52
Description: as for outcome 4
Time Frame: Baseline, Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 14 | 17 | 29 | 35
Score on a scale | -0.804 (0.3099) | -0.885 (0.2962) | -0.773 (0.3374) | -0.967 (0.3920)

21. Secondary Outcome: Part B: Change From Baseline in Mean Eosinophilic Esophagitis Histology Scoring System (EoE-HSS) Stage Score at Week 52
Description: as for outcome 5
Time Frame: Baseline, Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 14 | 17 | 29 | 35
Score on a scale | -0.767 (0.3114) | -0.855 (0.3485) | -0.784 (0.3183) | -0.892 (0.3181)

22. Secondary Outcome: Part B: Absolute Change From Baseline in EoE Endoscopic Reference Total Score (EoE-EREFS) at Week 52
Description: The EoE-EREFS is a validated endoscopic scoring system for inflammatory and remodeling features of EoE including edema, rings, exudates, furrows, and stricture. The score was assessed in the proximal and distal esophageal regions with each region scored from 0 to 9 with total scores possibly ranging from 0 to 18. Higher scores indicate worse endoscopic inflammatory and remodeling findings.
Time Frame: Baseline, Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 11 | 14 | 22 | 30
score on a scale | -5.82 (1.722) | -3.64 (3.342) | -4.50 (3.203) | -4.77 (3.081)

23. Secondary Outcome: Part B: Change From Baseline in the Proportion of Days With 1 or More EoE Signs Measured by Pediatric EoE Sign/Symptom Questionnaire - Caregiver Version (PESQ-C) at Week 52
Description: PESQ-C is a novel, observer-reported outcome measure intended to be completed independently by caregivers of all pediatric EoE participants in the study.
Time Frame: Baseline, Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 6 | 9 | 18 | 27
proportion of days | -0.20 (0.373) | -0.47 (0.395) | -0.49 (0.339) | -0.30 (0.299)

24. Secondary Outcome: Part B: Number of Sign-free Days During the 14-day Period Preceding Week 52 as Measured by the PESQ-C (for Participants Aged ≥1 to <12 Years)
Description: as for outcome 23
Time Frame: Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: sign-free days
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 6 | 9 | 18 | 27
sign-free days | 11.58 (3.968) | 12.10 (4.652) | 11.35 (3.947) | 12.13 (4.053)

25. Secondary Outcome: Part B: Change From Baseline in the Proportion of Total Segments Within a Day (Night, Morning, Afternoon, Evening) With 1 or More EoE Signs as Measured by the PESQ-C at Week 52
Description: PESQ-C is a novel, observer-reported outcome measure intended to be completed independently by caregivers of all pediatric EoE participants in the study. The PESQ-C measured the occurrence of signs of EoE and was completed once daily via an electronic diary.
Time Frame: Baseline, Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: proportion of segments
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 6 | 9 | 18 | 27
proportion of segments | -0.03 (0.249) | -0.24 (0.221) | -0.26 (0.250) | -0.17 (0.187)

26. Secondary Outcome: Part B: Change From Baseline in the Proportion of Days With 1 or More EoE Signs by Pediatric EoE Sign/Symptom Questionnaire - Participant Version (PESQ-P) (for Participants Aged ≥8 to <12 Years) at Week 52
Description: as for outcome 12
Time Frame: Baseline, Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 3 | 6 | 11 | 12
proportion of days | -0.33 (0.322) | -0.43 (0.369) | -0.42 (0.400) | -0.26 (0.396)

27. Secondary Outcome: Part B: Number of Symptom-free Days During the 14-day Period Preceding Week 52 as Measured by the PESQ-P (for Participants Aged ≥8 to <12 Years)
Description: The PESQ-P was a participant-reported outcome measure intended to be completed independently by participants ≥8 to <12 years of age. The PESQ-P measures the signs of EoE, including stomach pain, heartburn, acid reflux, regurgitation, vomiting, food refusal, and trouble swallowing food.
Time Frame: Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: sign-free days
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 3 | 6 | 11 | 12
sign-free days | 9.33 (8.083) | 11.67 (5.715) | 10.64 (4.943) | 13.63 (0.874)

28. Secondary Outcome: Part B: Change From Baseline in the Proportion of Total Segments Within a Day (Night, Morning, Afternoon, Evening) With 1 or More EoE Signs as Measured by the PESQ-P (for Participants Aged ≥8 to <12 Years) at Week 52
Description: as for outcome 14
Time Frame: Baseline, Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: proportion of segments
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 3 | 6 | 11 | 12
proportion of segments | -0.17 (0.164) | -0.26 (0.269) | -0.21 (0.293) | -0.16 (0.284)

29. Secondary Outcome: Part B: Normalized Enrichment Score (NES) for the Relative Change From Baseline in the EoE Diagnostic Panel (EDP) at Week 52
Description: A Normalized Enrichment Score (NES) is a way to generate a single numerical value to represent a complex gene expression signature. Changes in NES score represented the overall changes in the expression of that molecular phenotype. The NESs calculated for the EDP reflect the expression at post-baseline relative to Baseline of a gene set that is differentially expressed between esophageal biopsies from EoE participants compared to healthy controls as a way to evaluate normalization of the molecular pathology. For each subject, an NES of 0 indicates no change from baseline, a negative score shows a reduction in disease score (more like normal) and positive score shows worsening (more active disease). NES does not have minimum/maximum score.
Time Frame: Baseline, Week 52
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 8 | 12 | 16 | 21
Score on a scale | -2.715 [-2.755 to -2.505] | -2.615 [-2.810 to -2.430] | -2.625 [-2.775 to -2.550] | -2.670 [-2.710 to -2.530]

30. Secondary Outcome: Part B: Normalized Enrichment Score (NES) for the Relative Change From Baseline in the Type 2 Inflammation Signature (T2INF) at Week 52
Description: A Normalized Enrichment Score (NES) is a way to generate a single numerical value to represent a complex gene expression signature. Changes in NES score represented the overall changes in the expression of that molecular phenotype. The NESs calculated for T2INF reflect the expression at post-baseline relative to Baseline of the pre-specified gene set as a way to evaluate normalization of type 2 inflammation with treatment. For each subject, an NES of 0 indicates no change from baseline, a negative score shows a reduction in disease score (more like normal) and positive score shows worsening (more active disease). NES does not have minimum/maximum score.
Time Frame: Baseline, Week 52
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 8 | 12 | 16 | 21
Score on a scale | -1.960 [-2.000 to -1.895] | -1.965 [-1.995 to -1.765] | -1.920 [-1.965 to -1.865] | -1.920 [-1.930 to -1.850]

31. Secondary Outcome: Part B: Change From Baseline in Body Weight for Age Percentile at Week 52
Description: Body weight for age percentile was calculated based on the growth charts from the Centers for Disease Control and Prevention (CDC) for ages 0 to 20 years (for ages 2 to <12 years) and World Health Organization (WHO) growth charts for ages 0 to <2 years (for ages 1 to <2 years). These charts included a set of smoothed percentiles along with CDC LMS (Lambda-Mu-Sigma) parameters to allow the calculation of percentiles.
Time Frame: Baseline, Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percentile
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 14 | 16 | 29 | 35
Percentile | -0.02 (13.893) | 5.48 (12.644) | 4.75 (11.968) | 5.96 (11.519)

32. Secondary Outcome: Part B: Change From Baseline in Body Mass Index (BMI) for Age Z-score for Participants ≥2 Years of Age at Week 52
Description: BMI for age z-score indicates how much higher or lower a participant's BMI for age is relative to a reference growth chart (based on the growth charts from Centers for Disease Control and Prevention [CDC] for ages 0 to 20 years [for ages 2 to <12 years]). A z-score of "0" represents the population mean. An increase in the mean change in BMI for age z-score (ie, increase in the standard deviation [SD] from the reference growth chart) indicates an increase in BMI for age relative to the reference.
Time Frame: Baseline, Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 14 | 15 | 27 | 32
z-score | -0.0206 (0.54625) | 0.0687 (0.47605) | -0.0549 (0.88582) | 0.0987 (0.72329)

33. Secondary Outcome: Part B: Change From Baseline in Weight for Age Z-score at Week 52
Description: Weight for age z-score indicates how much higher or lower a participant's weight for age is relative to a reference growth chart (based on the growth charts from CDC for ages 0 to 20 years [for ages 2 to <12 years] and World Health Organization (WHO) growth charts for ages 0 to <2 years [for ages 1 to <2 years]). A z-score of "0" represents the population mean. An increase in the mean change in weight for age z-score (increase in the SD from the reference growth chart) indicates an increase in weight for age relative to the reference.
Time Frame: Baseline, Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 14 | 16 | 29 | 35
z-score | 0.0640 (0.46264) | 0.2016 (0.39446) | 0.1445 (0.40310) | 0.2049 (0.40305)

34. Secondary Outcome: Part B: Change From Baseline in Body Weight From Height Z-score at Week 52
Description: Weight for height z-score indicates how much higher or lower a participant's weight for height is relative to a reference growth chart (based on the growth charts from CDC for ages 0 to 20 years [for ages 2 to <12 years] and WHO growth charts for ages 0 to <2 years [for ages 1 to <2 years]). A z-score of "0" represents the population mean. An increase in the mean change in weight for height z-score (increase in the SD from the reference growth chart) indicates an increase in weight for height relative to the reference.
Time Frame: Baseline, Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 2 | 3 | 9 | 12
z-score | 0.0962 (0.48902) | -0.0100 (0.51706) | -0.2700 (1.04895) | -0.0151 (0.67968)

35. Secondary Outcome: Part B: Concentration of Functional Dupilumab in Serum at Week 32 and 52
Description: Concentration of functional dupilumab in serum at Week 32 and 52 was reported in this outcome measure.
Time Frame: Week 32 and 52
Population: Analysis was performed on PKAS. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 14 | 18 | 29 | 37
mg/L
  Week 32: number analyzed (Participants) | 13 | 17 | 28 | 36
  Week 32 | 105 (49.8) | 142 (48.5) | 99.0 (42.8) | 186 (59.5)
  Week 52: number analyzed (Participants) | 13 | 15 | 24 | 30
  Week 52 | 101 (44.3) | 149 (59.1) | 83.0 (33.2) | 179 (75.3)

36. Secondary Outcome: Part A: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, Adverse Events of Special Interest (AESIs) and TEAEs Leading to Permanent Discontinuation of Study Drug
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation patient administered with a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. A serious AE was any untoward medical occurrence that at any dose resulted in death, life-threatening, initial or prolonged inpatient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or a medically important event. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. TEAEs include both Serious TEAEs and non-serious TEAEs. An AESI was defined as one of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor was appropriate.
Time Frame: From Baseline up to Week 16 in Part A
Population: Analysis was performed on Part A SAF which included all randomized patients who received any Part A study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 34 | 37 | 30
Participants
  Participants with any TEAE | 31 | 27 | 26
  Participants with any Serious TEAE | 0 | 2 | 1
  Participants with any AESI | 1 | 2 | 1
  Participants with any TEAE leading to permanent discontinuation of study drug | 2 | 0 | 0

37. Secondary Outcome: Part B: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, Adverse Events of Special Interest (AESIs) and TEAEs Leading to Permanent Discontinuation of Study Drug
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation patient administered with a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. A serious AE was any untoward medical occurrence that at any dose resulted in death, life-threatening, initial or prolonged inpatient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or a medically important event. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. TEAEs include both Serious TEAEs and non-serious TEAEs. An AESI was defined as one of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor was appropriate.
Time Frame: From Week 16 up to Week 52 in Part B
Population: Analysis was performed on Part B SAF which included all participants who received at least 1 dose of Part B study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 14 | 18 | 29 | 37
Participants
  Participants with any TEAE | 14 | 15 | 28 | 34
  Participants with any Serious TEAE | 1 | 0 | 3 | 2
  Participants with any AESI | 0 | 1 | 3 | 4
  Participants with any TEAE leading to permanent discontinuation of study drug | 0 | 0 | 0 | 1

38. Secondary Outcome: Part A: Number of Participants With Positive Treatment-emergent Antidrug Antibodies (ADA) Response
Description: Treatment-emergent ADA was defined as a negative result or missing result at baseline with at least one positive post baseline result in the ADA assay. Samples positive in the dupilumab ADA assay were characterized for ADA titers (low, moderate and high). The low treatment-emergent ADA titer as defined as titer level <1000, moderate as 1000 to 10000 and high as >10000.
Time Frame: From Baseline up to Week 16 in Part A
Population: Analysis was performed on ADA analysis set (AAS) which included all participants who received any amount of study drug (active or placebo) and had at least one non-missing anti-drug antibody result following the first dose of study drug or placebo. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 25 | 31 | 26
Participants | 1 | 1 | 0

39. Secondary Outcome: Part A: Number of Participants With Positive Treatment-emergent Antidrug Antibodies (ADA) by Maximum Titer Category
Description: as for outcome 38
Time Frame: From Baseline up to Week 16 in Part A
Population: Analysis was performed on AAS which included all participants who received any amount of study drug (active or placebo) and had at least one non-missing anti-drug antibody result following the first dose of study drug or placebo. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and overall number of participants analyzed = 0 denotes that no participant had positive treatment-emergent ADA response to measure titer level.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Pooled Placebo | Part A: Dupilumab High Dose | Part A: Dupilumab Low Dose
Number analyzed (Participants) | 1 | 1 | 0
Participants
  Treatment-emergent ADA Titer: Low | 1 | 1 | 0
  Treatment-emergent ADA Titer: Moderate | 0 | 0 | 0
  Treatment-emergent ADA Titer: High | 0 | 0 | 0

40. Secondary Outcome: Part B: Number of Participants With Positive Treatment-emergent Antidrug Antibodies (ADA) Response and Titer
Description: Treatment-emergent ADA was defined as a negative result or missing result at baseline with at least one positive post baseline result in the ADA assay. Samples positive in the dupilumab ADA assay were characterized for ADA titers (low, moderate and high). The low treatment-emergent ADA titer as defined as titer level <1000, moderate as 1000 to 10000 and high as >10000.
  No participant exhibited a treatment-emergent ADA response in Part B and titer was not reported.
Time Frame: From Week 16 up to Week 52 in Part B
Population: Analysis was performed on AAS which included all participants who received any amount of study drug and had at least one non-missing anti-drug antibody result following the first dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo to Dupilumab Low Dose | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose
Number analyzed (Participants) | 14 | 18 | 29 | 37
Participants | 0 | 0 | 0 | 0

41. Secondary Outcome: Part C: Percentage of Participants Achieving Peak Esophageal Intraepithelial Eosinophil Count of <15 Eos/Hpf At Week 100
Time Frame: At Week 100
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Number; unit: Percentage of participants
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 41
Percentage of participants | 92.7

42. Secondary Outcome: Part C: Percentage of Participants Achieving Peak Esophageal Intraepithelial Eosinophil Count of <15 Eos/Hpf At Week 160
Time Frame: At Week 160
Population: No data was collected for this endpoint. No participants reached end of part C treatment period (week 160).
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 0

43. Secondary Outcome: Part C: Percent Change in Peak Esophageal Intraepithelial Eosinophil Count (Eos/Hpf) From Baseline to Week 100
Time Frame: Baseline to Week 100
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 41
Percentage of change | -91.50 (13.348)

44. Secondary Outcome: Part C: Percent Change in Peak Esophageal Intraepithelial Eosinophil Count (Eos/Hpf) From Baseline to Week 160
Time Frame: Baseline to Week 160
Population: No data was collected for this endpoint. No participants reached end of part C treatment period (week 160).
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 0

45. Secondary Outcome: Part C: Absolute Change in Mean EoE-HSS From Baseline to Week 100
Time Frame: Baseline to Week 100
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 41
Score on a scale
  EoE-HSS Grade Score | -0.851 (0.3909)
  EoE-HSS Stage Score | -0.850 (0.3648)

46. Secondary Outcome: Part C: Absolute Change in Mean EoE-HSS From Baseline to Week 160
Time Frame: Baseline to Week 160
Population: No data was collected for this endpoint. No participants reached end of part C treatment period (week 160).
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 0

47. Secondary Outcome: Part C: Absolute Change in EoE-EREFS From Baseline to Week 100
Time Frame: Baseline to Week 100
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 32
Score on a scale | -5.34 (2.535)

48. Secondary Outcome: Part C: Absolute Change in EoE-EREFS From Baseline to Week 160
Time Frame: Baseline to Week 160
Population: No data was collected for this endpoint. No participants reached end of part C treatment period (week 160).
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 0

49. Secondary Outcome: Part C: Change in Total Score as Measured by the PEESSv2.0- Caregiver Version Questionnaire From Baseline to Week 100
Description: The PEESSv2.0-C is a caregiver-reported outcome measure that assesses the frequency and severity of EoE symptoms among pediatric participants. The PEESSv2.0-C consists of 20 items and has a one-month recall period. Each item had a 0-4 scale, which was transformed to 0-100 as follows: 0 = 0, 1 = 25, 2 = 50, 3 = 75, 4 = 100. The mean total PEESSv2.0 score was computed as the sum of all the item scores over the number of items answered. The total PEESSv2.0-C score ranges from 0 to 100 where higher scores indicate greater symptom burden among pediatric EoE participants.
Time Frame: Baseline to Week 100
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 43
Score on a scale | -25.03 (21.867)

50. Secondary Outcome: Part C: NES for the Relative Change in the EDP Transcriptome Signature From Baseline to Week 100
Description: as for outcome 29
Time Frame: Baseline to Week 100
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 39
Score on a scale | -2.720 [-2.800 to -2.510]

51. Secondary Outcome: Part C: NES for the Relative Change in the EDP Transcriptome Signature From Baseline to Week 160
Description: as for outcome 29
Time Frame: Baseline to Week 160
Population: No data was collected for this endpoint. No participants reached end of part C treatment period (week 160).
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 0

52. Secondary Outcome: Part C: NES for the Relative Change in the Type 2 Inflammation Transcriptome Signature Baseline to Week 100
Time Frame: Baseline to Week 100
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 39
Score on a scale | -1.970 [-2.000 to -1.900]

53. Secondary Outcome: Part C: NES for the Relative Change in the Type 2 Inflammation Transcriptome Signature From Baseline to Week 160
Time Frame: Baseline to Week 160
Population: No data was collected for this endpoint. No participants reached end of part C treatment period (week 160).
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 0

54. Secondary Outcome: Part C: Change in Body Weight for Age Percentile From Baseline up to Week 100
Description: as for outcome 31
Time Frame: Baseline up to Week 100
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Mean (Standard Deviation); unit: Percentile
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 46
Percentile | 10.63 (18.227)

55. Secondary Outcome: Part C: Change in Body Mass Index for Age Z-score From Baseline up to Week 100
Description: Difference in the 100-week change from baseline in BMI-for-age Z-score. BMI-for-age Z-scores are based on a reference growth chart (based on the growth charts from Centers for Disease Control and Prevention [CDC] for ages 0 to 20 years [for ages 2 to <12 years]. A z-score of "0" represents the population mean. The Z-score indicates the number of standard deviations away from the mean of the reference population. A negative Z-score indicates values lower than the population mean while a positive Z-score indicates values higher than the population mean.
Time Frame: Baseline up to Week 100
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 45
z-score | 0.2009 (0.67389)

56. Secondary Outcome: Part C: Change in Weight for Age Z-score From Baseline up to Week 100
Description: Difference in the 100-week change from baseline in weight-for-age Z-score. Weight-for-age Z-scores are based on a reference growth chart (based on the growth charts from Centers for Disease Control and Prevention [CDC] for ages 0 to 20 years [for ages 2 to <12 years]. A z-score of "0" represents the population mean. The Z-score indicates the number of standard deviations away from the mean of the reference population. A negative Z-score indicates values lower than the population mean while a positive Z-score indicates values higher than the population mean.
Time Frame: Baseline up to Week 100
Population: Here 'n' = number of evaluable participants at the specified timepoint.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 46
z-score | 0.3376 (0.59272)

57. Secondary Outcome: Part C: Change in Weight for Age Z-score From Baseline up to Week 160
Description: Weight for age z-score indicates how much higher or lower a participant's weight for age is relative to a reference growth chart (based on the growth charts from CDC for ages 0 to 20 years [for ages 2 to <12 years] and World Health Organization (WHO) growth charts for ages 0 to <2 years [for ages 1 to <2 years]). An increase in the mean change in weight for age z-score (increase in the SD from the reference growth chart) indicates an increase in weight for age relative to the reference.
Time Frame: Baseline up to Week 160
Population: No data was collected for this endpoint. No participants reached end of part C treatment period (week 160).
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 0

58. Secondary Outcome: Part C: Change in Weight for Height Z-score From Baseline up to Week 100
Description: Difference in the 100-week change from baseline in Weight for height Z-score. Weight for height Z-scores are based on a reference growth chart (based on the growth charts from Centers for Disease Control and Prevention [CDC] for ages 0 to 20 years [for ages 2 to <12 years]. A z-score of "0" represents the population mean. The Z-score indicates the number of standard deviations away from the mean of the reference population. A negative Z-score indicates values lower than the population mean while a positive Z-score indicates values higher than the population mean.
Time Frame: Baseline up to Week 100
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 15
z-score | 0.3301 (0.84791)

59. Secondary Outcome: Part C: Change in Weight for Height Z-score From Baseline up to Week 160
Description: Weight for height z-score indicates how much higher or lower a participant's weight for height is relative to a reference growth chart (based on the growth charts from CDC for ages 0 to 20 years [for ages 2 to <12 years] and WHO growth charts for ages 0 to <2 years [for ages 1 to <2 years]). An increase in the mean change in weight for height z-score (increase in the SD from the reference growth chart) indicates an increase in weight for height relative to the reference.
Time Frame: Baseline up to Week 160
Population: No data was collected for this endpoint. No participants reached end of part C treatment period (week 160).
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 0

60. Secondary Outcome: Part C: Percentage of Participants Achieving Peak Esophageal Intraepithelial Eosinophil Count of ≤6 Eos/Hpf (400×) at Week 100
Time Frame: At Week 100
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Number; unit: Percentage of participants
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 41
Percentage of participants | 70.7

61. Secondary Outcome: Part C: Percentage of Participants Achieving Peak Esophageal Intraepithelial Eosinophil Count of ≤6 Eos/Hpf (400×) at Week 160
Time Frame: At Week 160
Population: No data was collected for this endpoint. No participants reached end of part C treatment period (week 160).
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 0

62. Secondary Outcome: Part C: Percentage of Participants (With Food Elimination Diet Regimens at Baseline) That Have a Re-introduction of a Previously Eliminated Food Group From Baseline up to Week 100
Time Frame: Baseline up to Week 100
Measure: Number; unit: Percentage of participants
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 61
Percentage of participants | 14.8

63. Secondary Outcome: Part C: Percentage of Participants (With Food Elimination Diet Regimens at Baseline) That Have a Re-introduction of a Previously Eliminated Food Group From Baseline up to Week 160
Time Frame: Baseline up to Week 160
Population: No data was collected for this endpoint. No participants reached end of part C treatment period (week 160).
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 0

64. Secondary Outcome: Part C: Number of Participants With TEAEs
Time Frame: Up to Week 152
Population: No participants completed 160 weeks, longest duration was 152 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 61
Participants | 53

65. Secondary Outcome: Part C: Number of Participants With Treatment-emergent SAEs
Time Frame: Up to Week 152
Population: No participants completed 160 weeks, longest duration was 152 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 61
Participants | 3

66. Secondary Outcome: Part C: Number of Participants With Treatment-emergent AESIs
Time Frame: Up to Week 152
Population: No participants completed 160 weeks, longest duration was 152 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 61
Participants | 6

67. Secondary Outcome: Part C: Number of Participants With TEAEs Leading to Permanent Discontinuation of Study Treatment
Time Frame: Up to Week 152
Population: No participants completed 160 weeks, longest duration was 152 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 61
Participants | 0

68. Secondary Outcome: Part C: Number of Participants With Treatment-emergent ADA Responses
Time Frame: From Week 52 up to Week 152
Population: Anti-Drug Antibody Analysis Set (AAS): The Part C AAS included all participants who received any amount of study drug in Part C and had at least 1 non-missing ADA result following the first dose of study drug. Analysis was based on treatment received.
Measure: Number; unit: Participants
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 39
Participants | 0

69. Secondary Outcome: Part C: Concentration of Functional Dupilumab in Serum at Week 100
Time Frame: At Week 100
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Part C: Dupilumab
Number analyzed (Participants) | 42
mg/L | 180 (96.9)

ADVERSE EVENTS:
Time Frame: From signing of the informed consent up to week 152.
Groups:
- Part B: Placebo to Dupilumab Low Dos: Participants who received subcutaneous (SC) injection of placebo in Part A and received lower exposure dupilumab in Part B. Lower exposure dupilumab regimen were exposures approximating those in adolescents and adults receiving 300 mg dupilumab Q2W
Arm/Group | Part A: Pooled Placebo (Placebo) | Part A: Dupilumab Low Dose | Part A: Dupilumab High Dose | Part B: Placebo to Dupilumab Low Dos | Part B: Placebo to Dupilumab High Dose | Part B: Dupilumab Low Dose to Dupilumab Low Dose | Part B: Dupilumab High Dose to Dupilumab High Dose | Part C: Dupilumab
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/30 | 0/37 | 0/14 | 0/18 | 0/29 | 0/37 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/30 | 2/37 | 1/14 | 0/18 | 2/29 | 2/37 | 3/61
Other Adverse Events (participants affected / at risk) | 28/34 | 24/30 | 26/37 | 14/14 | 16/18 | 27/29 | 31/37 | 48/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Pooled Placebo (Placebo) (N=34) | Part A: Dupilumab Low Dose (N=30) | Part A: Dupilumab High Dose (N=37) | Part B: Placebo to Dupilumab Low Dos (N=14) | Part B: Placebo to Dupilumab High Dose (N=18) | Part B: Dupilumab Low Dose to Dupilumab Low Dose (N=29) | Part B: Dupilumab High Dose to Dupilumab High Dose (N=37) | Part C: Dupilumab (N=61)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HCoV-OC43 infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal food impaction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endoscopy gastrointestinal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Pooled Placebo (Placebo) (N=34) | Part A: Dupilumab Low Dose (N=30) | Part A: Dupilumab High Dose (N=37) | Part B: Placebo to Dupilumab Low Dos (N=14) | Part B: Placebo to Dupilumab High Dose (N=18) | Part B: Dupilumab Low Dose to Dupilumab Low Dose (N=29) | Part B: Dupilumab High Dose to Dupilumab High Dose (N=37) | Part C: Dupilumab (N=61)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 8 (9) | 2 (2) | 8 (8)
Ear infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 5 (5)
Molluscum contagiosum (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (6) | 4 (4)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 3 (4)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 5 (7)
COVID-19 (Infections and infestations) | 0 (0) | 9 (9) | 6 (6) | 3 (3) | 6 (7) | 7 (7) | 11 (11) | 5 (6)
Vomiting (Gastrointestinal disorders) | 6 (15) | 1 (1) | 3 (7) | 0 (0) | 2 (2) | 3 (6) | 5 (7) | 11 (24)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 3 (3) | 4 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (2) | 1 (2) | 3 (9) | 3 (3) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 5 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (3) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 2 (3)
Injection site reaction (General disorders) | 7 (8) | 4 (11) | 4 (11) | 4 (34) | 5 (21) | 4 (17) | 5 (18) | 5 (32)
Injection site erythema (General disorders) | 1 (1) | 1 (2) | 4 (8) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 2 (4) | 3 (3) | 6 (7) | 11 (18)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (6) | 1 (1) | 1 (3) | 1 (1) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (2) | 1 (1) | 5 (7) | 4 (4) | 5 (6) | 8 (11)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 3 (4) | 2 (4) | 2 (4) | 1 (2) | 4 (7) | 5 (5)
Eczema (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (3) | 3 (3) | 0 (0) | 2 (2) | 1 (2) | 2 (2)
Seasonal allergy (Immune system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 4 (5)
Dizziness (Nervous system disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 4 (5) | 2 (2) | 0 (0) | 4 (4) | 3 (5) | 4 (4) | 6 (9)
Fear of injection (Psychiatric disorders) | 2 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (4) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Respiratory tract infection viral (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 1 (1) | 1 (1) | 2 (2)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 4 (5)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Ear infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Groin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 4 (4) | 4 (4) | 3 (3)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (4)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 2 (2) | 0 (0) | 13 (15)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 3 (3) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (3) | 6 (6)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 3 (4)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Oropharyngeal cobble stone mucosa (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 1 (2) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Enuresis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Immunisation reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (3) | 4 (4)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Gas poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Genital pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/51/NCT04394351/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/51/NCT04394351/SAP_002.pdf